CLINICAL TRIAL: NCT00974727
Title: Use of Biomarkers to Assess Unhealthy Lifestyle Contributions to Summer Weight Gain in Children
Brief Title: A Gardening Program to Assess Unhealthy Lifestyle Contributions to Summer Weight Gain in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MSN106189
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2009-09

CONDITIONS: Overweight
Keywords: Childhood overweight; Gardening; Summer weight gain
MeSH Terms: conditions — Overweight; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gardening Program (Experimental)
  Interventions: Other: Garden Fit
- Control (No Intervention): Subjects received the standard of care for the summer.

INTERVENTIONS:
Other: Garden Fit — 8-week summer gardening program. 9am-12pm on Monday, Wednesday, Friday and 9am-12:30pm on Tuesday and Thursday. Activities included gardening (preparing soil for planting, planting seeds and seedlings, mulching, weeding, watering, and harvesting), preparing meals with fresh foods from the garden, and other garden activities and games.
  Other Names: Garden Fit 2009
  Arms: Gardening Program

SUMMARY:
The purpose of this study is to examine the impact of a summer gardening program on summer weight gain in overweight middle school children.

DETAILED DESCRIPTION:
In the past two decades, the combination of unhealthy eating and physical inactivity has contributed to doubling the percentage of children and adolescents who are overweight. Childhood overweight is known to lead to increased risk for several morbidities in childhood and into adulthood including type 2 diabetes mellitus, hypertension, and cardiovascular disease. Recent data shows that children experience greater and more variable increases in BMI during summer vacation than during the school year. Our project aims to determine whether summer weight gain is due to a decrease in physical activity or an increase in daily calories as well as to assess the effectiveness of a summer gardening program on preventing summer body fat gain. We will randomize 40 middle-school children who are above the 95th percentile for BMI into either a control or intervention group. The control group will receive the standard of care and the intervention group will participate in Garden Fit, a summer gardening project at Troy Gardens in Madison, WI. As part of Garden Fit, subjects will participate in weeding, landscaping and trail maintenance activities as well as preparing meals twice a week with fresh foods from the gardens. We hypothesize that summer weight gain is due to a worsening of healthy lifestyle (decreased physical activity from school to summer and increased eating of high calorie snacks). Additionally, we hypothesize that an intervention that increases physical activity and provides increased access to healthy foods will reduce the trend of summer BMI increase.

ELIGIBILITY:
Inclusion Criteria:

* Middle school child aged 10-14 years
* BMI at or above the 85th percentile for height and weight
* Able to attend 8-week summer program and clinic visits

Exclusion Criteria:

* Any known metabolic disorder
* Any physical disability that prevents or limits physical activity
* Claustrophobia

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2009-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
BMI | June 2009 and August 2009

SECONDARY OUTCOMES:
Fitness (as measured by VO2 Submax testing) | June 2009 and August 2009
Resting Metabolic Rate | June 2009 and August 2009
Fasting insulin | June 2009 and August 2009
Fasting glucose | June 2009 and August 2009
CRP | June 2009 and August 2009
IL-6 | June 2009 and August 2009
Body Composition | June 2009 and August 2009
Plasma Carotenoids | June 2009 and August 2009
Total Energy Expenditure | June 2009 and August 2009
Food Consumption (measured by FFQs) | June 2009 and August 2009

CONTACTS AND LOCATIONS:
Overall Officials: Dale Schoeller, Ph.D., Principal Investigator — University of Wisconsin, Department of Nutritional Sciences
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

REFERENCES:
- [Background] Ogden CL, Flegal KM, Carroll MD, Johnson CL. Prevalence and trends in overweight among US children and adolescents, 1999-2000. JAMA. 2002 Oct 9;288(14):1728-32. doi: 10.1001/jama.288.14.1728. PMID 12365956
- [Background] Ferraro KF, Thorpe RJ Jr, Wilkinson JA. The life course of severe obesity: does childhood overweight matter? J Gerontol B Psychol Sci Soc Sci. 2003 Mar;58(2):S110-9. doi: 10.1093/geronb/58.2.s110. PMID 12646600
- [Background] Carrel AL, Clark RR, Peterson S, Eickhoff J, Allen DB. School-based fitness changes are lost during the summer vacation. Arch Pediatr Adolesc Med. 2007 Jun;161(6):561-4. doi: 10.1001/archpedi.161.6.561. PMID 17548760
- [Background] Gillis L, McDowell M, Bar-Or O. Relationship between summer vacation weight gain and lack of success in a pediatric weight control program. Eat Behav. 2005 Feb;6(2):137-43. doi: 10.1016/j.eatbeh.2004.08.002. PMID 15598600
- [Background] von Hippel PT, Powell B, Downey DB, Rowland NJ. The effect of school on overweight in childhood: gain in body mass index during the school year and during summer vacation. Am J Public Health. 2007 Apr;97(4):696-702. doi: 10.2105/AJPH.2005.080754. Epub 2007 Feb 28. PMID 17329660
- [Background] Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA. 2006 Apr 5;295(13):1549-55. doi: 10.1001/jama.295.13.1549. PMID 16595758
- [Background] Whitaker RC, Wright JA, Pepe MS, Seidel KD, Dietz WH. Predicting obesity in young adulthood from childhood and parental obesity. N Engl J Med. 1997 Sep 25;337(13):869-73. doi: 10.1056/NEJM199709253371301. PMID 9302300
- [Background] Hull HR, Morrow ML, Heesch KC, Dinger MK, Han JL, Fields DA. Effect of the summer months on body weight and composition in college women. J Womens Health (Larchmt). 2007 Dec;16(10):1510-5. doi: 10.1089/jwh.2006.0329. PMID 18062766
- [Background] Gutin B. Child obesity can be reduced with vigorous activity rather than restriction of energy intake. Obesity (Silver Spring). 2008 Oct;16(10):2193-6. doi: 10.1038/oby.2008.348. No abstract available. PMID 18719647
- [Background] Gutin B, Barbeau P, Owens S, Lemmon CR, Bauman M, Allison J, Kang HS, Litaker MS. Effects of exercise intensity on cardiovascular fitness, total body composition, and visceral adiposity of obese adolescents. Am J Clin Nutr. 2002 May;75(5):818-26. doi: 10.1093/ajcn/75.5.818. PMID 11976154
- [Background] Johnson L, Mander AP, Jones LR, Emmett PM, Jebb SA. Energy-dense, low-fiber, high-fat dietary pattern is associated with increased fatness in childhood. Am J Clin Nutr. 2008 Apr;87(4):846-54. doi: 10.1093/ajcn/87.4.846. PMID 18400706
- [Background] Wang YC, Bleich SN, Gortmaker SL. Increasing caloric contribution from sugar-sweetened beverages and 100% fruit juices among US children and adolescents, 1988-2004. Pediatrics. 2008 Jun;121(6):e1604-14. doi: 10.1542/peds.2007-2834. PMID 18519465
- [Background] Carrel AL, Clark RR, Peterson SE, Nemeth BA, Sullivan J, Allen DB. Improvement of fitness, body composition, and insulin sensitivity in overweight children in a school-based exercise program: a randomized, controlled study. Arch Pediatr Adolesc Med. 2005 Oct;159(10):963-8. doi: 10.1001/archpedi.159.10.963. PMID 16203942